CLINICAL TRIAL: NCT00749918
Title: Improved Insulin Sensitivity With Therapeutic Vitamin D Replacement in Pre-Diabetic Vitamin D Deficient Individuals
Brief Title: Effect of Vitamin D Deficiency and Vitamin D Supplementation on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin Healthcare Research Institute (Other)
Responsible Party: Shaban Nazarian, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0609M92006
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Prediabetes; Vitamin D Deficiency
Keywords: vitamin D; Cholecalciferol; Insulin sensitivity; MinMod Millennium; FSIGT; modified frequently sampled IV glucose tolerance test
MeSH Terms: conditions — Prediabetic State; Vitamin D Deficiency; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Each subject was evaluated and data was collected before and after the intervention
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (vitamin D3) — Oral capsules of cholecalciferol, 5000 IU/ capsule, two capsules daily for one month.
  Other Names: Cholecalciferol by BIO-TECH Pharmacal, Inc.

SUMMARY:
This study was intended to evaluate the effect of vitamin D supplementation on insulin sensitivity and pancreatic islet beta-cell function. Our hypothesis was that vitamin D supplementation to normal levels in patients with impaired fasting glucose will result in improved insulin sensitivity and improved beta cell function.

DETAILED DESCRIPTION:
A modified frequently sampled intravenous glucose tolerance (mFSIGT) test was used. On day 0, baseline 22 time point mFSIGT was performed. Subjects were then treated with cholecalciferol (vitamin D3) supplementation - 10,000 IU/day - for 28 consecutive days. mFSIGT was then repeated measuring glucose, insulin and c-peptide at all time points. 25-OH vitamin D, PTH, and calcium were also measured at time point 0 pre and post vitamin D supplementation. Data was analyzed using the Bergman/Boston minimal model for insulin homeostasis with MinMod Millennium software.

ELIGIBILITY:
Inclusion Criteria:

* Impaired fasting glucose
* Adult, age between 18 and 65
* Serum vitamin D level below 30 ng/mL

Exclusion Criteria:

* History of nephrolithiasis
* Any medications that can effect insulin sensitivity or beta cell function (i.e. antipsychotics, metformin)
* Pregnancy
* Liver disease
* Renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Assessment of insulin sensitivity before and after oral vitamin D3 supplementation with 10,000 IU/day for one month. | At baseline and after 4 weeks of vitamin D supplementation

SECONDARY OUTCOMES:
Monitor effect of vitamin D supplementation with 10,000 IU/day for one month on serum calcium and parathyroid hormone levels. | One month
Assess effect of vitamin D supplementation on beta cell function as measured by analysis of data collected through a modified FSIGT test. | One month

CONTACTS AND LOCATIONS:
Overall Officials: Cary Mariash, MD, Study Director — University of Minnesota; Shaban Nazarian, MD, Principal Investigator — University of Minnesota; Sidney Jones, MD, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota, Division of Endocrinology, Minneapolis, Minnesota, United States